CLINICAL TRIAL: NCT02094183
Title: The Interaction Between Appetite Hormones and Their Importance for Maintenance of Weight Loss After a Low Calorie Diet
Brief Title: The Interaction Between Appetite Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Principal Investigator, Signe Torekov, Assistant professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-4-2010-134
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucagon-Like Peptide 1; Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 (Experimental): GLP-1 and low calorie diet
  Interventions: Other: GLP-1; Dietary Supplement: low calorie diet
- Control (Experimental): low calorie diet
  Interventions: Dietary Supplement: low calorie diet

INTERVENTIONS:
Other: GLP-1 — GLP-1
  Arms: GLP-1
Dietary Supplement: low calorie diet — low calorie diet

SUMMARY:
Glucagon Like Peptide (GLP) -1 affects metabolic response corrected for weight change

DETAILED DESCRIPTION:
Many obese people have had several successful weight losses, however very few can maintain the weight loss over a longer period (e.g. one year) Therefore, we want to investigate the metabolic response and the importance for maintenance of weight loss in obese people, who lost at least 7, 5 % body weight by low calorie diet followed by 52 weeks of diet weight maintenance with or without supplement of GLP-1.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 and < 40 (kg/m2)
* Healthy

Exclusion Criteria:

* Other known illness
* Medicine that affects glucose- and lipid metabolism, appetite or food intake
* Pregnancy
* Breast feeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in hormone level corrected for weight change | Baseline and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Jens Holst, DMSCi, Study Chair — University of Copenhagen
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen
  - Hvidovre University Hospital, Hvidovre

REFERENCES:
- [Derived] Brethvad AO, Zakariassen HL, Holt J, Lundgren JR, Jakobsen A, Hartmann B, Lehmann EW, Kissow H, Holst JJ, Madsbad S, Torekov SS, Holst B. Increased meal-induced neurotensin response predicts successful maintenance of weight loss - Data from a randomized controlled trial. Metabolism. 2023 Jun;143:155534. doi: 10.1016/j.metabol.2023.155534. Epub 2023 Mar 16. PMID 36933790
- [Derived] Akawi N, Checa A, Antonopoulos AS, Akoumianakis I, Daskalaki E, Kotanidis CP, Kondo H, Lee K, Yesilyurt D, Badi I, Polkinghorne M, Akbar N, Lundgren J, Chuaiphichai S, Choudhury R, Neubauer S, Channon KM, Torekov SS, Wheelock CE, Antoniades C. Fat-Secreted Ceramides Regulate Vascular Redox State and Influence Outcomes in Patients With Cardiovascular Disease. J Am Coll Cardiol. 2021 May 25;77(20):2494-2513. doi: 10.1016/j.jacc.2021.03.314. PMID 34016263
- [Derived] Iepsen EW, Lundgren JR, Hartmann B, Pedersen O, Hansen T, Jorgensen NR, Jensen JE, Holst JJ, Madsbad S, Torekov SS. GLP-1 Receptor Agonist Treatment Increases Bone Formation and Prevents Bone Loss in Weight-Reduced Obese Women. J Clin Endocrinol Metab. 2015 Aug;100(8):2909-17. doi: 10.1210/jc.2015-1176. Epub 2015 Jun 4. PMID 26043228